CLINICAL TRIAL: NCT04577560
Title: Does the Telomere Length in First Human Polar Body Correlates With the Telomere Length in Cumulus Cells: A Clinical Validation Study
Brief Title: Telomere Length in Human Polar Body and Telomere Length in Cumulus Cells: A Clinical Validation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Ana Arnanz, Principal Investigator, ART Fertility Clinics LLC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-ABU-007-AA
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Telomere Length
Keywords: PGT-A; telomere length; cumulus cells; polar body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MII with PB biopsy (Experimental): Five selected MII will undergo sequential polar biopsy; on day 0 [PB1] (36-42 hours post trigger injection) and if fertilization occurred on day 1 [PB2] (17-20 hours post ICSI). On day 5, 6 or 7, the resulting blastocyst will be biopsied.
  Interventions: Genetic: First polar body biopsy in MII oocytes; Genetic: PGT-A blastocyst
- MII with no PB biopsy (Experimental): MII will not go under polar body biopsy. On day 5, 6 or 7, the resulting blastocyst will be biopsied.
  Interventions: Genetic: PGT-A blastocyst

INTERVENTIONS:
Genetic: First polar body biopsy in MII oocytes — Since PBs are by-products of the meiotic division of the oocyte and are not required for fertilization and subsequent embryo development, they can be removed to assess exclusively maternal chromosomal information without harming the embryo integrity. As previously described, PB biopsy does not impact the morphokinetic parameters of the embryo development and can be safely applied without the risk of impairing the reproductive potential of the embryo.
  Other Names: telomere lenght
  Arms: MII with PB biopsy
Genetic: PGT-A blastocyst — preimplantation genetic screening for aneuploidies

SUMMARY:
To investigate whether telomere length (TL) of the first Polar body (PB) correlates with TL in Cumulus cells (CC)

DETAILED DESCRIPTION:
With the present study we want to analyze, as a primary objective, whether telomere length (TL) in the first Polar Body (PB) correlates with TL in the corresponding Cumulus cells (CC). As a secondary objective, a possible correlation between TL in PBs and blastocyst TL and ploidy will be evaluated.

To our best knowledge, there are no studies evaluating TL in CC and TL in PBs of the corresponding oocyte. With the present prospective study, we sought to investigate whether there is a correlation between CC-TL and PB-TL. If a correlation exists, CC-TL assessment would serve as a valuable non-invasive technique to gain information about oocyte competence.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18- 30kg/m2
* Expected normo/high responders
* Normal female/male karyotype
* Antagonist protocol with agonist trigger.
* PGT-A: NGS in blastocysts
* Fresh autologous ejaculates (≥5 mill/ml)
* Primary and secondary infertility
* Only ICSI as insemination technique

Exclusion Criteria:

• PCOS patients according to International evidence-based guideline for the assessment and management of polycystic ovarian syndrome 2018.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
telomere length (TL) of the first Polar body (PB) and TL in Cumulus cells (CC) | 8 weeks
  Correlation between telomere length (TL) of the first Polar body (PB) and TL in Cumulus cells (CC)

SECONDARY OUTCOMES:
To correlate TL between both polar bodies | 8 weeks
  If the MII fertilize after performing ICSI, polar body biopsy for the second PB will be performed
To correlate TL in male WBC and TL in sperm | 8 weeks
  TL will be assess in leukocytes (male´s blood sample) and in the sperm (fresh ejaculate)
To correlate TL in female WBC and TL in CC | 8 weeks
  TL will be assess in leukocytes (female´s blood sample) and in the cumulus cells (CC) from the retrieved oocytes.
To evaluate a possible correlation between TL-CC and TL-TE | 8 weeks
  Correlation between TL-CC and TL in trophectoderm biopsy performed in the developed blastocysts
To evaluate a possible correlation between TL-CC and ploidy TE | 8 weeks
  Correlation between TL-CC and PGT-A results in trophectoderm biopsy performed in the developed blastocysts
To evaluate telomerase activity (TA) in CC and a possible correlation with CC-TL | 8 weeks
  Telomerase is a ribonucleoprotein complex responsible for de novo telomere synthesis and addition of telomeric repeats to existing telomeres
To evaluate FSH/LH gene expression in CC | 8 weeks
  During the follicular phase LH whose receptors (LHR) are expressed in granulosa cells under the influence of FSH, plays an important role in the regulation of ovarian function and is essential to promote the growth of the dominant follicle, final oocyte maturation as well as ovulation induction
To evaluate a possible correlation between ploidy in PBs and ploidy in TE biopsy | 8 weeks
  PGT-A in PB and PGT-A in TE biopsy
PB biopsy and embryo development | 8 weeks
  To validate that PB biopsy does not impair embryo development compared to their sibling embryos with no PB biopsied
To evaluate TL in sperm + TL-PB and TL in TE | 8 weeks
  TL in sperm + TL-PB and TL in the resulting biopsied

CONTACTS AND LOCATIONS:
Overall Officials: Ana Arnanz Poyatos, MSc, Principal Investigator — ART Fertility Clinics
Locations (1):
- ART Fertility Clinics, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: From March 2021
Access Criteria: pubmed
URL: https://pubmed.ncbi.nlm.nih.gov

REFERENCES:
- [Result] Kosebent EG, Uysal F, Ozturk S. Telomere length and telomerase activity during folliculogenesis in mammals. J Reprod Dev. 2018 Dec 14;64(6):477-484. doi: 10.1262/jrd.2018-076. Epub 2018 Sep 28. PMID 30270279
- [Result] Ozturk S. Telomerase activity and telomere length in male germ cells. Biol Reprod. 2015 Feb;92(2):53. doi: 10.1095/biolreprod.114.124008. Epub 2015 Jan 7. PMID 25568305
- [Result] Riethman H, Ambrosini A, Paul S. Human subtelomere structure and variation. Chromosome Res. 2005;13(5):505-15. doi: 10.1007/s10577-005-0998-1. PMID 16132815
- [Result] Keefe DL, Marquard K, Liu L. The telomere theory of reproductive senescence in women. Curr Opin Obstet Gynecol. 2006 Jun;18(3):280-5. doi: 10.1097/01.gco.0000193019.05686.49. PMID 16735827
- [Result] Kidder GM, Vanderhyden BC. Bidirectional communication between oocytes and follicle cells: ensuring oocyte developmental competence. Can J Physiol Pharmacol. 2010 Apr;88(4):399-413. doi: 10.1139/y10-009. PMID 20555408
- [Result] Cheng EH, Chen SU, Lee TH, Pai YP, Huang LS, Huang CC, Lee MS. Evaluation of telomere length in cumulus cells as a potential biomarker of oocyte and embryo quality. Hum Reprod. 2013 Apr;28(4):929-36. doi: 10.1093/humrep/det004. Epub 2013 Feb 1. PMID 23377770
- [Result] Lara-Molina EE, Franasiak JM, Marin D, Tao X, Diaz-Gimeno P, Florensa M, Martin M, Seli E, Pellicer A. Cumulus cells have longer telomeres than leukocytes in reproductive-age women. Fertil Steril. 2020 Jan;113(1):217-223. doi: 10.1016/j.fertnstert.2019.08.089. Epub 2019 Oct 6. PMID 31594634
- [Result] Wang W, Chen H, Li R, Ouyang N, Chen J, Huang L, Mai M, Zhang N, Zhang Q, Yang D. Telomerase activity is more significant for predicting the outcome of IVF treatment than telomere length in granulosa cells. Reproduction. 2014 Apr 8;147(5):649-57. doi: 10.1530/REP-13-0223. Print 2014 May. PMID 24472817
- [Result] Montag M, Koster M, Strowitzki T, Toth B. Polar body biopsy. Fertil Steril. 2013 Sep;100(3):603-7. doi: 10.1016/j.fertnstert.2013.05.053. Epub 2013 Jun 21. PMID 23796365
- [Result] Treff NR, Su J, Taylor D, Scott RT Jr. Telomere DNA deficiency is associated with development of human embryonic aneuploidy. PLoS Genet. 2011 Jun;7(6):e1002161. doi: 10.1371/journal.pgen.1002161. Epub 2011 Jun 30. PMID 21738493
- [Result] Schenk M, Groselj-Strele A, Eberhard K, Feldmeier E, Kastelic D, Cerk S, Weiss G. Impact of polar body biopsy on embryo morphokinetics-back to the roots in preimplantation genetic testing? J Assist Reprod Genet. 2018 Aug;35(8):1521-1528. doi: 10.1007/s10815-018-1207-4. Epub 2018 May 22. PMID 29790071